CLINICAL TRIAL: NCT00636779
Title: BraveNet Multi-Center Integrative Medicine Survey
Brief Title: BraveNet Integrative Medicine Descriptive Study
Acronym: BraveNet
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: The Bravewell Collaborative (Other); Alliance Institute for Integrative Medicine (Other); Allina Health System (Other); Scripps Center for Integrative Medicine (Other); University of California, San Francisco (Other); University of Maryland (Other); The Continuum Center for Health and Healing (Unknown); Thomas Jefferson University (Other); Venice Family Clinic (Other)
Responsible Party: Rowena Dolor, Coordinating Principal Investigator, Bravewell Integrative Medicine Research Network (BraveNet)
Other Study IDs: Pro00006850
Record Dates: First submitted 2008-03-09; First posted 2008-03-14 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2011-06

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Up to five hundred eligible patients seen at each of the nine participating Integrative Medicine Centers will be approached (by mail, phone, at the time of their visit, etc.) and invited to consent to the paper and pencil study.

SUMMARY:
The Bravewell Integrative Medicine Research Network (BraveNet) is a newly formed practice-based research network of nine leading integrative medicine centers around the U.S. collaborating in clinical outcomes research to increase the knowledge and evidence-base of integrative medicine.

DETAILED DESCRIPTION:
Specific Aims of BraveNet:

1. Demonstrate feasibility for the nine sites of BraveNet to coordinate in specifying data elements, developing and implementing smooth data collection procedures, analyzing the data, publishing and disseminating the results through scientific conferences and journals.
2. Describe the patients seeking care at Integrative Medicine centers, in terms of:

   1. demographics, presenting symptoms, health conditions, type of care sought, and expectations for treatment;
   2. quality of life, mood, stress; and
   3. lifestyle factors.
3. Explore potential patterns within the sample [e.g., do the survey scores vary by demographics, by condition, by type patient (new vs return), by type of help sought, etc.].
4. Utilize above data as pilot data for future studies and funding opportunities.

Up to five hundred eligible patients seen at each of the nine participating Centers will be approached (by mail, phone, at the time of their visit, etc.) and invited to consent to the paper and pencil study. The patient survey will clearly state that participation is voluntary with a written consent to participate on the front. Individual practices will report the response rate in order to monitor the potential effect of volunteer bias. Participant completion of questionnaires should take 15 to 30 minutes, and should be completed within 2 weeks of the patient visit., The corresponding provider form will be completed by the provider/research staff within 5 days of the visit.

Measures:

1. Baseline Questionnaires - Demographics and reason for visit
2. Quality of Life. The SF-12 (Short Form 12)
3. Mood (Depression). The Center for Epidemiologic Studies Depression Scale (CES-D)
4. Stress. The Perceived Stress Scale (PSS)
5. Visual Analog Scales (VAS). Four self-report VASs will be used to measure aspects of pain, fatigue and restfulness of sleep.
6. Provider Form. Providers/ Research Staff will complete this form to indicate the type of provider seen, the CPT codes used to describe/bill for the service, the services provided, and the provider's assessment of current medical conditions/co-morbidities.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible for inclusion in this study only if all of the following criteria apply:

  1. Age: At least 18 years of age.
  2. Patient Status: Participants are eligible if seen individually by any type of clinician on the day of the visit.
  3. English or Spanish Literacy: Ability to read and write English or Spanish as confirmed by the site personnel and ability to provide informed consent.

Exclusion Criteria:

* Subjects will be excluded from this study if any of the following criteria apply:

  1. Cognitive Impairment: A subject will not be eligible if he/she has a history of psychiatric disease, dementia, Alzheimer's disease, or other conditions which will limit the validity of providing informed consent to participate in the study.
  2. Inability to read and write in English or Spanish.
  3. Participating only in educational Center activities, not as a clinical patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 500 patients from each of the nine participating Integrative Medicine Centers who are seeing any type of clinicial on the day of their visit.
Sampling Method: Non-Probability Sample
Enrollment: 4340 (Actual)
Dates: Start 2008-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Describe the patients seeking care at Integrative Medicine centers, in terms of:a.demographics, presenting symptoms, health conditions, type of care sought, and expectations for treatment; b.quality of life, mood, stress; and c.lifestyle factors. | Once per patient

SECONDARY OUTCOMES:
Explore potential patterns within the sample [e.g., do the survey scores vary by demographics, by condition, by type patient (new vs return), by type of help sought, etc.]and utilize data as pilot data for future studies and funding opportunities. | Once all surveys have been entered into the EDC system

CONTACTS AND LOCATIONS:
Overall Officials: Rowena Dolor, MD, Principal Investigator — Duke Clinical Research Institute; Ruth Wolever, PhD, Principal Investigator — Duke Integrative Medicine Center
Locations (8):
- United States (8):
  - Scripps Center for Integrative Medicine, La Jolla, California
  - Osher Center for Integrative Medicine, San Francisco, California
  - Venice Family Clinic, Santa Monica, California
  - University of Maryland Center for Integrative Medicine, Baltimore, Maryland
  - Penny George Institute for Health and Healing, Minneapolis, Minnesota
  - Duke Integrative Medicine, Durham, North Carolina
  - Alliance Center for Integrative Medicine, Cincinnati, Ohio
  - Jefferson-Myrna Brind Center of Integrative Medicine, Philadelphia, Pennsylvania